## **Informed Consent Form**



## Cover page

Official title: Study protocol for a Randomised Controlled trial of Dance-movement Therapy for Adolescents with Depression

Date of the document: 6. December 2025

Registration details: This study is registrated at Clinical Trails, identifier HUS391/2021 NCT ID not yet assigned



Informed Consent form Version 2 6.12.2025

## CONSENT FOR PARTICIPATION IN RESEARCH

| Dance-movement therapy for adolescent depress<br>HUS Psychiatry, adolescent outpatient unit | sion |
|---|---|
| I have been requested to gather information on the benefits of dance-movement therap | participate aforementioned scientific research to by in the treatment of depression. |
| I have read and understood the research information handout the provided guidelines. I have received sufficient informationing and handling out data. The information of patient record information of diagnostic interviews, measurements about we tion and level of education. The contents of the information handout have been communicanswers for all of my questions. Information was received from I have had adequate time to consider my participation. I have pose and practice of the research, including the benefits, risks persuasion to participate. | n about the research including the collection, process-<br>will be collected, such as visits to doctor and nurse,<br>ell-being, diagnoses, medical treatments, living condi-<br>icated to me orally and I have received<br>in the personnel of the adolescent outpatient unit.<br>he received sufficient information regarding the pur- |
| I know that the data will be processed confidentially and will not be disclosed to outsiders. I understand that participating the research is voluntary. I acknowledge that I have a right to refuse participation. I can discontinue participation and withdraw my consent at any time without providing a reason, and this will not affect my treatment in any way. | |
| I acknowledge that if I discontinue the research or withdraw my consent, the information obtained up to that point may still be utilized as a part of the research. | |
| I understand that expenses incurred form participating in the study will not be reimbursed. Caretaker is informed about the research by mail. Date: | |
| I confirm participation to this research and provide vo | luntary consent by signature. |
| Signature of the examinee | Date |
| Print name of the examinee | Date of birth of the examinee |
| Address of the examinee | - |

| Consent received | |
|------------------------------|------|
| Researcher / nurse signature | Date |
| Print name | |

The original signed document will be retained in the research files and a copy of the signed document will be provided to the examinee.